CLINICAL TRIAL: NCT05876624
Title: High Stakes, High Pressure: The Connection Between Personality, Burnout, and Hypertension in Nigerian Bank Employees
Brief Title: The Connection Between Personality, Burnout, and Hypertension in Nigerian Bank Employees
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Renaissance University Ugbawka, Enugu (Other)
Responsible Party: Principal Investigator, Lawrence Ugwu, Researcher, Renaissance University Ugbawka, Enugu
Other Study IDs: RenaissanceU
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood Pressure measurement — Blood Pressure measurement
  Other Names: Blood Pressure

SUMMARY:
This is a longitudinal study which we plan to examine the link between personality traits, burnout, and hypertension in bank employees in South-eastern Nigeria

DETAILED DESCRIPTION:
This proposed longitudinal study aims to examine the relationship between personality traits, burnout, and hypertension in bank employees in South-eastern Nigeria, where hypertension is a significant public health issue. The study will involve bankers as participants, who will be asked to complete self-report questionnaires and measure their blood pressure over four weeks. The research seeks to determine if personality differences and burnout levels contribute to hypertension risk in this population. By understanding the role of psychosocial factors in hypertension risk, the study hopes to provide recommendations for workplace adjustments that could improve employee well-being and reduce hypertension risk among Nigerian bank employees.

ELIGIBILITY:
Inclusion Criteria:

* Any staff of the Bank

Exclusion Criteria:

* Non Staff

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all Staff of commercial banks in Nigeria
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-05-22 (Estimated); Primary Completion 2023-06-19 (Estimated); Study Completion 2023-07-10 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 20 minutes
  Blood Pressure measurement

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence E Ugwu, Principal Investigator — Renaissance University Ugbawka Enugu Nigeria
Locations (1):
- Renaissance University, Enugu, Nigeria

IPD SHARING:
Plan to Share IPD: No
We No plan of sharing the data.